CLINICAL TRIAL: NCT05879263
Title: "Efficacy of Intermittent Enteral Nutrition Versus Continuous Administration in Intensive Care Patients for the Reduction of Complications. Randomized Clinical Trial"
Brief Title: "Efficacy of Intermittent Enteral Nutrition Versus Continuous Administration in Intensive Care"
Acronym: ENINCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Complejo Hospitalario Universitario de Albacete (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Maria Dolores Saiz Vinuesa, Principal Investigator, Complejo Hospitalario Universitario de Albacete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUA_59_07_2021
Record Dates: First submitted 2023-05-03; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Enteral Nutrition; Critical Care; Feeding Methods; Gastric Feeding Tube
Keywords: Gastric Emptying; Diarrea; Vomiting; Respiratory Aspiration of Gastric Content; Caloric Intake; Enteral nutrition; Critical care
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Intervention Model Description: The patients wil be allocated to expriemental group or control group using a simple randomization sequence.
  There is an allocation concealment using sealed opaque envelopes Duration: From February 2022 to complete sample number.
Masking Description: By the nature of the intervention(intermittent or continuous administration of enteral nutrition) is impossible to mask it to participats, care provider or investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERMITTENT ENTERAL NUTRITITION (IEN) (Experimental): Administration of Enteral Nutriton (EN) by nasogastric tube in 4 bolus (24h): Duration of the infusion 1hour each shot, using an infusion pump.
  Interventions: Other: INTERMITTENT ENTERAL NUTRITITION (IEN)
- CONTINUOUS ENTERAL NUTRITION (CEN) (Active Comparator): Administration of Enteral Nutriton (EN) by nasogastric tube during 24 hours, using an infusion pump.
  Interventions: Other: CONTINUOS ENTERAL NUTRITITION (CEN)

INTERVENTIONS:
Other: INTERMITTENT ENTERAL NUTRITITION (IEN) — Administration of Enteral Nutriton (EN) by nasogastric tube in 4 bolus (24h): Duration of the infusion 1hour each shot, using an infusion pump.
  Arms: INTERMITTENT ENTERAL NUTRITITION (IEN)
Other: CONTINUOS ENTERAL NUTRITITION (CEN) — Administration of Enteral Nutriton (EN) by nasogastric tube during 24 hours, using an infusion pump.
  Arms: CONTINUOUS ENTERAL NUTRITION (CEN)

SUMMARY:
The goal of this clinical trial is to Determine efficacy of intermittent enteral nutrition vs continuous enteral nutrition in adults patients with a nasogastric tube in a intensive care unit.

The main question[s] it aims to answer are:

* Reduction of gastrointestinal and respiratory complications
* Evaluate the achievement of the caloric objective Informed consent will be requested from participants who meet the inclusion criteria.

The participants will be randomized into two groups: control group (continuous enteral nutrition) or experimental group (intermittent enteral nutrition) Researchers will compare intermittent enteral nutrition vs continuous to see if there is a reduction in gastrointestinal and respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU of University General Hospital of Albacete
* Need for enteral nutrition by nasogastric tube in the first 48 hours
* Signed informed consent

Exclusion Criteria:

* Insulin dependent diabetic patients
* Abdominal surgery
* Dire prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory Complications | during ICU stay (maximum 15 days)
  Respiratory aspiration of gastric content
Gastrointestinal Complications | during ICU stay (maximum 15 days)
  Digestive intolerance: Diarrhea, vomiting, increased gastric residual volume(GRV)

SECONDARY OUTCOMES:
Achievement of the caloric objective | during ICU stay (up to 15 days)
  Time in hours to reach caloric goal
Nutritional status: MNA | up to two days after admission to the ICU
  Measure with:Mini Nutritional Assessment,(MNA) 12-14 points: Normal nutritional status 8-11 points: risk of malnutrition 0-7 points: Malnutrition
Changes in blood glucose | during ICU stay (maximum 15 days)
  Episodes of hypoglycemia or hyperglycemia
ICU Stay | From date of randomization until 100 months
  Days of stay in ICU
Mortality | until the date of death from any cause until 100 months
  Percentage of deaths in ICU
Change of type of EN administration | during ICU stay (maximum 15 days)
  Change of EN administration modality
Nutritional status:Glim Criteria | up to two days after admission to the ICU
  Measure with: Glim criteria: Phenotypic criteria:Non-volitional weight loss (%) Low BMI (kg/m2)Reduced muscle mass(calf circumference (cm)) Etiologic criteria: Reduced food intake or assimilation. Inflammation
  *Requires at least one phenotypic criterion and one etiologic criterion for the diagnosis of malnutrition
Nutritional status: Biochemical values | up to two days after admission to the ICU
  Measure with:biochemical values: albumin, prealbumin, total protein

CONTACTS AND LOCATIONS:
Overall Officials: M.Dolores Saiz-Vinuesa, NURSE, Principal Investigator — Gerencia de Atención Integrada de Albacete
Locations (1):
- Maria Dolores Saiz Vinuesa, Albacete, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen YC. Critical analysis of the factors associated with enteral feeding in preventing VAP: a systematic review. J Chin Med Assoc. 2009 Apr;72(4):171-8. doi: 10.1016/S1726-4901(09)70049-8. PMID 19372071
- [Result] Lewis SR, Schofield-Robinson OJ, Alderson P, Smith AF. Enteral versus parenteral nutrition and enteral versus a combination of enteral and parenteral nutrition for adults in the intensive care unit. Cochrane Database Syst Rev. 2018 Jun 8;6(6):CD012276. doi: 10.1002/14651858.CD012276.pub2. PMID 29883514
- [Result] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Result] Patel JJ, Rosenthal MD, Heyland DK. Intermittent versus continuous feeding in critically ill adults. Curr Opin Clin Nutr Metab Care. 2018 Mar;21(2):116-120. doi: 10.1097/MCO.0000000000000447. PMID 29232262
- [Result] Tavares de Araujo VM, Gomes PC, Caporossi C. Enteral nutrition in critical patients; should the administration be continuous or intermittent? Nutr Hosp. 2014 Mar 1;29(3):563-7. doi: 10.3305/nh.2014.29.3.7169. PMID 24559000
- [Result] Serpa LF, Kimura M, Faintuch J, Ceconello I. Effects of continuous versus bolus infusion of enteral nutrition in critical patients. Rev Hosp Clin Fac Med Sao Paulo. 2003 Jan-Feb;58(1):9-14. doi: 10.1590/s0041-87812003000100003. Epub 2003 Apr 30. PMID 12754584
- [Result] Ichimaru S. Methods of Enteral Nutrition Administration in Critically Ill Patients: Continuous, Cyclic, Intermittent, and Bolus Feeding. Nutr Clin Pract. 2018 Dec;33(6):790-795. doi: 10.1002/ncp.10105. Epub 2018 Jun 20. PMID 29924423
- [Result] Thong D, Halim Z, Chia J, Chua F, Wong A. Systematic review and meta-analysis of the effectiveness of continuous vs intermittent enteral nutrition in critically ill adults. JPEN J Parenter Enteral Nutr. 2022 Aug;46(6):1243-1257. doi: 10.1002/jpen.2324. Epub 2022 Feb 13. PMID 34965317
- [Result] Heffernan AJ, Talekar C, Henain M, Purcell L, Palmer M, White H. Comparison of continuous versus intermittent enteral feeding in critically ill patients: a systematic review and meta-analysis. Crit Care. 2022 Oct 25;26(1):325. doi: 10.1186/s13054-022-04140-8. PMID 36284334
- See also: Effectiveness of continuous enteral nutrition versus intermittent enteral nutrition in intensive care patients: a systematic review. — http://www.joannabriggslibrary.org/jbilibrary/index.php/jbisrir/article/view/1129